CLINICAL TRIAL: NCT02009540
Title: Efficacy of Peri-trigonal Onabotulinumtoxin Injections in the Treatment of Refractory Idiopathic Detrusor Overactivity (IDO): A Single-blind, Randomised Controlled Trial Comparing Peri-trigonal Injections vs Injection of the Bladder Body.
Brief Title: Botulinum Toxin in the Treatment of Idiopathic Detrusor Overactivity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mr HD Flood (Other)
Responsible Party: Sponsor-Investigator, Mr HD Flood, Consultant Urologist, University Hospital of Limerick
Organization: University Hospital of Limerick (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UHL02/2013
Record Dates: First submitted 2013-11-29; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Overactive Detrusor
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin injected to bladder body (Placebo Comparator): arm will receive 100u of onaBoNT-A in 20x1ml aliquots (5u/ml). 20 injections will be given into the bladder wall, sparing the trigone. Injections will be given through all layers of the bladder eg suburothelially and intradetrusor.
  Interventions: Drug: Botulinum toxin injected to bladder body
- Botulinum toxin injected into trigone (Active Comparator): Arm B will receive 100u onaBoNT-A injected into 10x1ml suburothelial peri-trigonal sites (aliquot dose 10u/ml).
  Interventions: Drug: Botulinum toxin injected into trigone

INTERVENTIONS:
Drug: Botulinum toxin injected to bladder body — arm will receive 100u of onaBoNT-A in 20x1ml aliquots (5u/ml). 20 injections will be given into the bladder wall, sparing the trigone. Injections will be given through all layers of the bladder eg suburothelially and intradetrusor. The intervention will be performed under local anaesthetic using a flexible cystoscope.
  Other Names: Botulinum toxin; Onabotulinumtoxin; Botox
  Arms: Botulinum toxin injected to bladder body
Drug: Botulinum toxin injected into trigone — Arm B will receive 100u onaBoNT-A injected into 10x1ml suburothelial peri-trigonal sites (aliquot dose 10u/ml). The procedure will be performed under local anaesthetic by flexible cystoscopy.
  Other Names: Botulinum toxin; Onabotulinumtoxin; Botox
  Arms: Botulinum toxin injected into trigone

SUMMARY:
Overactive Bladder (OAB) is a chronic condition caused by instability of the detrusor or bladder muscle, which gives rise to symptoms of urinary urgency and often urinary incontinence. Idiopathic Detrusor Overactivity (IDO) is a subset of OAB where the cause for the bladder muscle instability is unknown.

OAB is usually treated by conservative measures or with oral medications eg. anticholinergics. Injection of onabotulinum toxin A (onaBoNT-A) into the bladder wall is licenced in the treatment of refractory IDO where oral medications fail. The injected toxin paralyses the bladder by blocking the ability of certain (motor) nerves to communicate with the bladder muscle. As these nerves are mainly concentrated in what is known as the "body" of the bladder this is traditionally where the injections are given.

In addition to its action on motor nerves, onaBoNT-A also affects sensory nerve pathways. Recent studies show that IDO is caused by both motor and sensory nerve dysfunction, therefore injecting the "trigone", a part of the bladder where sensory nerves are particularly dense, may be of clinical benefit. Three studies comparing trigone versus trigone-sparing injection of botulinum toxin in the treatment of IDO have been carried out. One of these indicated a significant benefit in targeting the trigone and the other two did not show any difference.

Our study aims to examine if injection of onaBoNT-A into the trigone alone will provide symptom and functional improvement in patients with IDO by comparing peritrigonal injection of onaBoNT-A with the traditional method of injection which spares the trigone.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil ICS criteria for OAB
* Urodynamically proven detrusor instability
* Symptoms lasting >6/12
* Patients must discontinue anticholinergic medication >14 days prior to randomisation and withhold the use of anticholinergics for the duration of the study.
* Patients with mixed incontinence are eligible if their urge symptoms are predominant. These will be instruced to record only episodes of urge urinary incontinence.
* Providing informed consent to participate in the study
* At least 18 years of age

Exclusion Criteria:

* Previous BoNT-A injection within 9 months of randomisation
* History of any neurological condition e.g. MS, Parkinsons, CVA
* Contraindication to BoNT e.g. Myaesthenia gravis
* Urinary tract infection in previous 6/12
* Antimicrobial therapy in previous 6/12
* Previous or current diagnosis of prostate or bladder cancer
* History of treatment with cyclophosphamide
* Radiation cystitis
* Urethral dilatation, cystometrogram, bladder cystoscopy under anaesthetic or a bladder biopsy in previous 3/12
* Augmentation cystoplasty, cystectomy or neurectomy
* Urethral stricture of <12ch
* Pregnancy
* Sexually active women of childbearing potential who are unwilling to use contraceptive measures for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Global Response Assessment | measured at 3 months following intervention

SECONDARY OUTCOMES:
Functional outcomes - 3 day sensation related bladder diary | measured at 3 months following intervention
  Three day sensation related bladder diary
IIQ-7 quality of life questionnaire | measured at 3 months following intervention
Treatment tolerability - numerical rating scale (0-10) | measured at 2 weeks following intervention
UDI-6 quality of life questionnaire | measured at 3 months following intervention

CONTACTS AND LOCATIONS:
Overall Officials: H D Flood, FRCSI, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital of Limerick, Limerick, Ireland